CLINICAL TRIAL: NCT01147419
Title: The Study to Compare the Treatment of Stent and Prothesis Bypass in SFA Occlusions
Brief Title: Comparison of Stent and Prothesis Bypass in Superficial Femoral Artery
Acronym: SPACIAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Liu Changwei, the department of vascular surgery of PUMCH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-vascular surgery
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Arterial Occlusive Diseases; Vascular Diseases
Keywords: critical limb ischemia; peripheral artery occlusive disease; femoropopliteal artery bypass; Stent
MeSH Terms: conditions — Arterial Occlusive Diseases; Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1 | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bypass (Experimental): Patients presenting with long occlusion of the superficial femoral artery enrolled in bypass arm will undergo suprageniculate femoropopliteal bypass surgery to bypass the occluded superficial femoral artery. And the graft will be artificial blood vessel.
  Interventions: Device: femoral-popliteal bypass with artificial blood vessel
- stent (Experimental)
  Interventions: Device: stent

INTERVENTIONS:
Device: stent — Before operation, take aspirin 100mg every day. During the operation, stent is delivered by a catheter and positioned through the narrowing in the artery. The stent is then expanded against the wall of the blood vessel to provide a wider channel for blood. At last, use balloon dilate the stent.
  Arms: stent
Device: femoral-popliteal bypass with artificial blood vessel — Before operation, take aspirin 100mg every day. Groin and suprageniculate incision, PTFE graft with end to side anastomoses.
  Arms: bypass

SUMMARY:
Different strategies exist in the treatment of chronic long occlusion of the superficial femoral artery. Traditionally, these patients should be treated with bypass. If the great saphenous vein is unavailable, doctor has to choose artificial vessel as graft. Now, the skill of endovascular treatment is developing rapidly, and lots of doctors think most of such patients could be treated with stent. The purpose of this trial is to compare stent and artificial blood vessel bypass in the treatment of long occlusion of the superficial femoral artery. The study hypothesis is that patency rates are comparable and therefore the minimal invasive treatment of stent can be considered in such patients.

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, controlled trial to compare the therapeutic effect of stent and artificial blood vessel bypass to chronic long occlusion of the superficial femoral artery. Totally 200 patients will be entered into the trial. The study population will consist of patients with long superficial femoral stenosis and occlusion lesion (≥15 cm), presenting symptomatic ischemia（Rutherford 3-6）. The lesion does not extend beyond the aortoiliac artery or blow-knee popliteal artery, with at least 1 vessel infra-popliteal runoff to the foot.

Trial participants will be randomized to either stent group or artificial blood vessel bypass group.

Patients will be followed up for 3 years. Study examinations will be done at screening, procedure time, 1, 6, 12, 24 and 36 months after procedure.

This study will be conducted at 3 centers in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

* The patients volunteer to join the trial and sign the formal consent.
* The patients are ≥45 year-old and ≤80 year-old.
* The patients suffer from symptomatic leg ischemia with rutherford classification3, 4 , 5 or 6. The presentation is severe intermittent claudication, rest pain, ulcer or gangrene.
* The total length of the femoral and popliteal artery lesion(including ≥75% stenosis and occlusion) are at least 15cm.
* The femoral-popliteal artery has never received bypass or endovascular therapy before.
* No obvious stenosis or occlusion in the aortoiliac artery; or the lesion could be treated simultaneously or has already been cured.
* No obvious stenosis in below-knee popliteal artery; at least 1 vessel infra-popliteal runoff to the foot.
* No surgical contraindications;no infection in operation region.
* No available saphenous vein.

Exclusion Criteria:

* Refuse random treatment.
* Previous operations on the superficial femoral artery.
* Acute lower extremity arterial thrombosis.
* Serious major organ failure.
* Allergic to the contrast agent or has contrast nephropathy.
* No clinical compliance or unfit to join the trial.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Occlusion of the stent or artificial blood vessel bypass | 36 months

SECONDARY OUTCOMES:
Mortality | 30 days
  The number of death during the first month after procedure, no matter whether the cause of death is related to the procedure.
Rate of limb salvage | 36 months
Procedural complications, defined as any adverse event | 36 months
  including MI, DVT, hematoma, renal failure, wound infection, lymphatic fistula
Quality of Life assessment | 36 months
  assessment in 1 month,6 months,12 months,24 months and 36 months post procedure
Rate of amputation | 36 months
Increase in Ankle Brachial Index | 36 months
Restenosis measured by Duplex Ultrasound or CTA | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Liu Changwei, bachelor, Study Chair; Ye Wei, doctor, Principal Investigator
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality

REFERENCES:
- See also: the website of the vascular surgery department of PUMCH — http://www.vascular.cn/